CLINICAL TRIAL: NCT05065164
Title: Attending Doctor of Shenzhen People's Hospital
Brief Title: Denosumab and Screw Fixation for Osteoporotic Compression Fracture
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: no partcipants enrolled
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ShenzhenPH spine wang02
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Denosumab Allergy
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dnosumab (Experimental): Desuzumab 60 mg subcutaneously /6 months, twice a year
  Interventions: Drug: Denosumab Only Product
- placebo control (Placebo Comparator): Placebo subcutaneous injection /6 months, twice a year
  Interventions: Drug: Denosumab Only Product

INTERVENTIONS:
Drug: Denosumab Only Product — denosumab subcutaneous injection /6 months, twice a year
  Other Names: Denosumab

SUMMARY:
Evaluation of bone mineral density and function at 1 year after screw internal fixation of osteoporotic vertebral compression fractures with desuzumab: a parallel double-blind randomized controlled clinical trial

DETAILED DESCRIPTION:
Conduct a single-center, double-blind, randomized controlled clinical trial according to clinical Trial Reporting Standards (CONSORT). Bone mineral density and function were compared 1 year after screw internal fixation of osteoporotic vertebral compression fracture (OVCF) with desomumab versus placebo in Shenzhen People's Hospital from September, 2021 to September, 2022. The study was approved by Shenzhen People's Hospital and informed consent was signed

ELIGIBILITY:
Inclusion Criteria:• Must be age between 40 and 90 years old

* X-ray diagnosis of 1-2 vertebral compression fractures
* Dual energy X ray test bone mineral density T value less than -1
* fracture history lasted within 6 weeks
* MRI showed bone marrow edema of injured segment
* lower back pain, local spines tenderness

Exclusion Criteria:

* • Must be able to have no posterior vertebral wall fracture

  * Must be able to have no patients with intervertebral fissure
  * Must be able to have no infection
  * Must be able to have no malignancy
  * Must be able to have no neurological dysfunction
  * Must be able to have no previous use of anti-osteoporosis drugs within 6 weeks
  * Must be able to have no inability to perform magnetic resonance imaging
  * Must be able to have no prior back surgery
  * Must be able to have no other established contraindications for elective surgery

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
age | up to 12 months
  participants age (year)
sex | up to 12 months
  participants sex
height | up to 12 months
  participants height cm
weight | up to 12 months
  participants weight kg
BMI | up to 12 months
  participants body mass index
osteocalcin | up to 12 months
  osteocalcin in the N terminal molecular fragment
Procollagen type 1 n-terminal propeptide P1NP | up to 12 months
  Procollagen type 1 n-terminal propeptide
C-terminal cross-linked type 1 collagen terminal peptide CTX | up to 12 months
  C-terminal cross-linked type 1 collagen terminal peptide
Serum total calcium | up to 12 months
  Serum total calcium level
parathyroid hormone | up to 12 months
  serum parathyroid hormone level
albumin | up to 12 months
  serum albumin level
lumber spine bone mineral density | up to 12 months
  Dual energy X-ray for lumber spine bone mineral density
Hip bone mineral density | up to 12 months
  Dual energy X-ray for hip bone mineral density
MRI of lumber | up to 12 months
  Bone marrow edema and adjacent intervertebral disc were detected by MRI
pain visual analogue scores (VAS) | up to 12 months
  pain visual analogue scores (VAS) use categories to differentiate pain intensity, with 0 being "painless" and 100 being "the worst pain imaginable".

SECONDARY OUTCOMES:
The Roland-Morris Disability Questionnaire | up to 12 month
  The Roland-Morris Disability Questionnaire is a health status measure designed to be completed by patients to assess physical disability due to low back pain.
QUALEFFO 31 | up to 12 month
  Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO) was developed in 1997 to evaluate quality of life for patients with osteoporosis
EuroQol-5D (EQ-5D): an instrument for measuring quality of life | up to 12 month
  EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Wang, Doctor, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- ShenzhenPH, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No